CLINICAL TRIAL: NCT04620707
Title: RGS@Home Project: Scaling ICT Based Neurorehabilitation to Personalized 24/7 Home Care Post-stroke
Brief Title: RGS@Home: Personalized 24/7 Home Care Post-stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Bioengineering of Catalonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGS@Home2020
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Hemiparesis;Poststroke/CVA; Stroke, Acute; Motor Disorders; Spasticity, Muscle
MeSH Terms: conditions — Stroke; Motor Disorders; Muscle Spasticity | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RGS based therapy (Experimental)
  Interventions: Device: RGS based training and monitoring
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Therapy as usual

INTERVENTIONS:
Device: RGS based training and monitoring — The RGS treatment will consist in a variable number of sessions per week of RGS-based training. Each session consists of cognitive and motor training involving reaching, grasping, placing virtual objects. The duration of the training period will be variable. Patients will use the RGS@Clinic from admission to discharge, and will have the RGS@Home during the first 3 months of the outpatient stage after recruitment. After this period of time, the patient will be evaluated by clinicians and the RGS@Home system will be collected. The RGS-Wear will be kept by the patient also during the follow-up period, up to 1 year post-recruitment.
  Arms: RGS based therapy
Behavioral: Therapy as usual — The patients will follow treatment as usual, including conventional rehabilitation and physical therapy when corresponding. The exact treatment that the patients will receive will depend on the local medical guidelines.
  Arms: Treatment as usual

SUMMARY:
Stroke represents one of the main causes of adult disability and will be one of the main contributors to the burden of disease in 2030. However, the healthcare systems are not able to respond to the current demand let alone its future increase. There is a need to deploy new approaches that advance current rehabilitation methods and enhance their efficiency.

One of the latest approaches used for the rehabilitation of a wide range of deficits of the nervous system is based on virtual reality (VR) applications, which combine training scenarios with dedicated interface devices. Market drivers exist for new ICT based treatment solutions. IBEC/ Eodyne Systems has developed and commercialised the Rehabilitation Gaming System (RGS), a science-based ICT solution for neurorehabilitation combining brain theory, AI, cloud computing and virtual reality and targeting motor and cognitive recovery after stroke. RGS provides a continuum of evaluations and therapeutic solutions that accompany the patient from the clinic to the therapy centre. RGS has been clinically validated showing its superiority over other products while reducing cost also through its use of standard off-the-shelf hardware and a Software as a Service model (SaaS). Commercial evaluations have shown that RGS acts as a workforce multiplier while delivering a high quality of care at clinical centres (RGS@Clinic). However, in order to achieve significant benefits in the patients' QoL, it is essential that RGS becomes an at home solution providing 24/7 monitoring and care. For this reason, this project aims at investigating the RGS acceptability and adoption model.

The findings derived from this study will contribute to establish a novel and superior neurorehabilitation paradigm that can accelerate the recovery of hemiparetic stroke patients. Besides the clinical impact, such achievement could have relevant socioeconomic impact.

ELIGIBILITY:
Inclusion criteria:

* Patients presenting a first-ever ischemic or intracerebral hemorrhagic stroke.
* A CT SCAN and/or MRI had exclude other pathologies.
* Lesion localization by clinical symptoms/signs.
* Moderate to mild proximal upper limb motor impairment (MRC≥2).
* Age 20-85 years old.
* Able to sit on a chair or a wheelchair interacting with the RGS during a full session, and be capable and willing to participate in RGS therapy.

Exclusion criteria:

* Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.
* Severe cognitive capabilities that prevent the execution of the experiment (MoCA < 19). This cut-off score is based on pilot study (Maier, M. et al, 2019).
* Arteriovenous malformation or lesions not related with a stroke.
* Severe associated impairment such as spasticity, communication disabilities (sensorial, Wernicke aphasia or apraxia), major pain or other neuromuscular impairments or orthopedic devices that would interfere with the correct execution of the experiment (Modified Ashworth Scale < 3).
* Unable to use the RGS independently according to the therapist's observations and lacking support from a caregiver to use the RGS.
* Refusal to sign the consent form.
* Pre-stroke history of upper limb motor disability.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in the score of the upper extremity section of the Fugl-Meyer Assessment Test [min=0, max=66]. Higher scores indicate better functioning. | 12 weeks.
  Change in score from baseline to end of treatment (12 weeks).

SECONDARY OUTCOMES:
Change in Barthel Index [min=0, max=100]. Higher scores indicate better functioning. | 12 weeks.
  Change in score from baseline to end of treatment (12 weeks).
Change in Barthel Index [min=0, max=100]. Higher scores indicate better functioning. | 12 months.
  Change in score from baseline to end of treatment (12 months).
Number of patients that are readmitted into the hospital (inpatient) after being discharged to at-home status. | 12 months.
  Number of patients from baseline to 12 months post-baseline.
Change in the Stroke Specific Quality Of Life scale (SS-QOL) [min=49, max=245]. Higher scores indicate better functioning. | 12 weeks.
  Change in score from baseline to end of treatment (12 weeks).
Change in the Stroke Specific Quality Of Life scale (SS-QOL) [min=49, max=245]. Higher scores indicate better functioning. | 12 months.
  Change in score from baseline to follow-up (12 months).
Change in the SIS (Stroke impact Scale) [min=0, max=42]. Higher scores indicate better functioning. | 12 weeks.
  Change in score from baseline to end of treatment (12 weeks).
Change in the SIS (Stroke impact Scale) [min=0, max=42]. Higher scores indicate better functioning. | 12 months.
  Change in score from baseline to follow-up (12 months).
Change in the Hamilton Scale Depression [min=0, max=52]. Lower scores indicate less impairment. | 12 weeks.
  Change in score from baseline to end of treatment (12 weeks).
Change in the Hamilton Scale Depression [min=0, max=52]. Lower scores indicate less impairment. | 12 months.
  Change in score from baseline to follow-up (12 months).
Change in the Visual Analogue Score (VAS) [min=0, max=10]. Lower scores indicate less impairment. | 12 weeks.
  Change in score from baseline to end of treatment (12 weeks).
Change in the Ashworth Scale [min=0, max=4]. Lower scores indicate less impairment. | 12 months.
  Change in score from baseline to follow-up (12 months).
Change in the Fatigue Severity Scale [min=9, max=63]. Higher scores indicate more fatigue. | 12 weeks.
  Change in score from baseline to end of treatment (12 weeks).
Change in the Fatigue Severity Scale [min=9, max=63]. Higher scores indicate more fatigue. | 12 months.
  Change in score from baseline to follow-up (12 months).
Change in the Wellbeing questionnaire (SF-36) [min=0, max=100]. Higher scores indicate more wellbeing. | 12 weeks.
  Change in score from baseline to end of treatment (12 weeks).
Change in the Wellbeing questionnaire (SF-36) [min=0, max=100]. Higher scores indicate more wellbeing. | 12 months.
  Change in score from baseline to follow-up (12 months).
Change in the score of the upper extremity section of the Fugl-Meyer Assessment Test. [min=0, max=66]. Higher scores indicate better functioning. | 12 months.
  Change in score from baseline to follow-up (12 months).

OTHER OUTCOMES:
Number of falls reported by the participants. | 12 weeks.
Number of falls reported by the participants. | 12 months.
Change in Barthel Index [min=0, max=100]. Higher scores indicate better functioning. | 6 months.
  Change in score from baseline to follow-up (6 months).
Change in the stroke specific Quality of Life scale (SS-QOL) [min=49, max=245]. Higher scores indicate better functioning. | 6 months.
  Change in score from baseline to follow-up (6 months).
Change in the Wellbeing questionnaire (SF-36) [min=0, max=100]. Higher scores indicate more wellbeing. | 6 months.
  Change in score from baseline to follow-up (6 months).
Change in the score of the upper extremity section of the Fugl-Meyer Assessment Test [min=0, max=66]. Higher scores indicate better functioning. | 6 months.
  Change in score from baseline to follow-up (6 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Bioengineering of Catalonia - Specs Lab, Barcelona, Spain

REFERENCES:
- [Derived] Mura A, Maier M, Ballester BR, De la Torre Costa J, Lopez-Luque J, Gelineau A, Mandigout S, Ghatan PH, Fiorillo R, Antenucci F, Coolen T, Chivite I, Callen A, Landais H, Gomez OI, Melero C, Brandi S, Domenech M, Daviet JC, Zucca R, Verschure PFMJ. Bringing rehabilitation home with an e-health platform to treat stroke patients: study protocol of a randomized clinical trial (RGS@home). Trials. 2022 Jun 20;23(1):518. doi: 10.1186/s13063-022-06444-0. PMID 35725616